CLINICAL TRIAL: NCT04705220
Title: Effect of Nutritional Supplementation With Turmeric on the Cognitive Performance of Subjects With Metabolic Syndrome
Acronym: EPICURO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indena S.p.A (Industry)
Collaborators: Istituto Superiore di Sanità (Other); Sintesi Research Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CUR-01-2019
Record Dates: First submitted 2019-12-06; First posted 2021-01-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment
Keywords: Metabolic Syndrome; Curcumin; Mild Cognitive Impairment; Nutraceutical; Nutritional Supplementation
MeSH Terms: conditions — Cognitive Dysfunction; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, single-center clinical trial. Patients enrolled will be randomized in a 1:1 ratio between groups and sexes to receive the test product MERIVA® (Group A) or its correspondent placebo (Group B).
Who Masked: Participant, Investigator
Masking Description: The test product MERIVA® is formulated in tablets indistinguishable from those of its correspondent placebo, with a completely indistinguishable appearance even in packaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Supplementation with Test Product (Experimental): Subjects will receive 1 tablet of MERIVA® in two administrations per day (one in the morning, one in the evening during meals) for a period of 6 months. This treatment corresponds to 1 g / day of experimental product (corresponding to about 200 mg of curcuminoids).
  Interventions: Dietary Supplement: MERIVA® Tablets
- Control Group without Nutritional Supplementation (Placebo Comparator): Subjects will receive 1 tablet of placebo in two administrations per day (one in the morning, one in the evening during meals) for a period of 6 months.
  Interventions: Other: Placebo Tablets

INTERVENTIONS:
Dietary Supplement: MERIVA® Tablets — The treatment corresponds to 1 g / day of experimental product (corresponding to about 200 mg of curcuminoids).
  Arms: Nutritional Supplementation with Test Product
Other: Placebo Tablets — The composition of placebo includes the same components of the treatment tablets, except for the active substance.
  Arms: Control Group without Nutritional Supplementation

SUMMARY:
The EPICURO study aims to demonstrate the beneficial effects of a 6-month dietary supplementation with an improved bioavailable turmeric (MERIVA®) on inflammatory, oxidative and metabolic parameters together with cognitive performance, potentially resulting in the reduction of the risk of cognitive decline in subjects, male and female, with Metabolic Syndrome. The results obtained will provide novel insights on MERIVA® for improving the prevention of age-related cognitive decline and Alzheimer's disease.

DETAILED DESCRIPTION:
This single-center trial will be a placebo-controlled, double-blind, randomized, 2 parallel groups study. The subjects will be randomly allocated to one of two treatment groups (MERIVA® or placebo). The duration of the supplementation is 6 months. The total sample size at baseline is 100 subjects aged 60+ years with Metabolic Syndrome, and therefore at risk of cognitive decline but without definite cognitive pathologies.

The primary objective of the study is the evaluation of the effect of nutritional supplementation with MERIVA® on the cognitive performance of subjects with Metabolic Syndrome, and therefore at risk of cognitive decline, with a view to maintaining the homeostatic balance of the function.

The secondary objectives of the study are:

* Evaluation of the effect of nutritional supplementation with turmeric (MERIVA®) on memory, executive and attention functions, language, neuropsychiatric profile and daily living ability of Subjects with Metabolic Syndrome;
* Evaluation of the effect of nutritional supplementation with turmeric (MERIVA®) on the body composition of Subjects with Metabolic Syndrome;
* Evaluation of the effect of nutritional supplementation with turmeric (MERIVA®) on the arterial properties of Subjects with Metabolic Syndrome;
* Evaluation of the effect of nutritional supplementation with turmeric (MERIVA®) on glucose metabolism and on the lipid and immune structure of Subjects with Metabolic Syndrome;
* Evaluation of the influence of gender / gender on the response to nutritional supplementation with turmeric (MERIVA®) in Subjects with Metabolic Syndrome;
* Confirmation of the safety profile of nutritional supplementation with turmeric (MERIVA®) in Subjects with Metabolic Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects.
* Subjects aged ≥ 60 years.
* Subjects with Metabolic Syndrome diagnosed according to standard criteria:

  1. Presence of abdominal obesity (waist circumference> 94 cm for males and> 80 cm for females).

     In addition, at least two of the following alterations:
  2. Fasting blood glucose ≥ 100 mg / dl.
  3. Triglycerides ≥ 150 mg / dl.
  4. HDL cholesterol <40 mg / dl for males, <50 mg / dl for females.
  5. Arterial hypertension (≥ 135/85 mmHg).
* Subjects who understand the nature of the study and provide their informed consent to participate.
* Subjects willing and able to participate in the visits and in the procedures foreseen by the study protocol.

Exclusion Criteria:

* Subjects with dementia with MMSE <24 test and on therapy with cholinesterase inhibitors or memantine*.
* Subjects with serious concomitant internal medical conditions or with neurological pathologies capable of causing cognitive dysfunction.
* Subjects with hepato-biliary disorders, including bile duct obstruction, cholangitis, gallstones.
* Subjects addicted to alcohol or drugs, or treated with psychotropic drugs at the time of enrollment.
* Subjects with known or suspected allergy or hypersensitivity to turmeric or other components of the experimental / placebo product.
* Subjects with Mild Cognitive Impairment (MCI) and in experimental therapy with Alzheimer's disease drugs.
* Subjects who are participating or have participated in other clinical studies within 30 days before enrollment.
* Subjects unable to sign the Informed Consent to Participation.

  * In case of conversion to dementia the Subjects will be kept in the study, will be subjected to the most appropriate therapies provided for the dementia pathology but will not enter the subsequent statistical evaluations.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Mini-Mental State Examination (MMSE) Test | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Percentage of subjects showing an improvement in performance in Mini-Mental State Examination (MMSE) test in comparison to baseline, defined as an increase of more than 2 points in the test. A difference between the group treated with MERIVA® versus placebo of at least 20% in the proportion of subjects with clinical improvement as defined above is considered clinically relevant. The differences between genders are considered.
Change from Baseline of Montreal Cognitive Assessment (MOCA) Test | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Percentage of subjects showing an improvement in performance in Montreal Cognitive Assessment (MOCA) test in comparison to baseline, defined as an increase of more than 2 points in the test. A difference between the group treated with MERIVA® versus placebo of at least 20% in the proportion of subjects with clinical improvement as defined above is considered clinically relevant. The differences between genders are considered.

SECONDARY OUTCOMES:
Change from Baseline of Rey's Auditory Verbal Learning Test (RAVLT) Test | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of the neuropsychological measurement performed regarding memory tests (Rey's Auditory Verbal Learning Test - RAVLT). Any differences between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.
Change from Baseline of Trail Making Test (TMT) Test | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of the neuropsychological measurement performed regarding executive functions and attention (Trail Making Test - TMT). Any differences between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.
Change from Baseline of Multiple Features Target Cancellation (MFTC) Test | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of the neuropsychological measurement performed regarding executive functions and attention (Multiple Features Target Cancellation - MFTC). Any differences between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.
Change from Baseline of Phonological and Semantic Verbal Fluidity (FVS) Test | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of the neuropsychological measurement performed regarding language (Phonological and Semantic Verbal Fluidity - FVS). Any differences between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.
Change from Baseline of Geriatric Depression Scale (GDS) Test | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of the neuropsychological measurement performed regarding a neuropsychiatric scale (Geriatric Depression Scale - GDS). Any differences between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.
Change from Baseline of Neuro-Psychiatric Inventory (NPI) Test | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of the neuropsychological measurement performed regarding a neuropsychiatric scale (Neuro-Psychiatric Inventory - NPI). Any differences between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.
Change from Baseline of Basic Activities of Daily Living (BADL) Test | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of the neuropsychological measurement performed regarding the ability to live everyday (Basic Activities of Daily Living - BADL). Any differences between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.
Change from Baseline of Instrumental Activities of Daily Living (IADL) Test | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of the neuropsychological measurement performed regarding the ability to live everyday (Instrumental Activities of Daily Living - IADL). Any differences between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.
Change from Baseline of Stroop Test - Short Version | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of the neuropsychological measurement performed regarding executive functions and attention (Stroop test short version). Any differences between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.
Change from Baseline of Bioelectrical Impedance (BIA) Assessment | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of body composition by bioelectrical impedance (BIA). Any differences between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.
Change from Baseline of Metabolism Parameters measured in Blood | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of metabolism changes (blood panel including: total cholesterol, Low-Density Lipoproteins, High-Density Lipoproteins, insulin, triglycerides, glucose, creatinine, uric acid, electrolytes, hepatic transaminases, gamma-glutamyltransferase, total proteins). In particular, any differences in terms of fasting blood glucose reduction and Homeostatic Model Assessment (HOMA) Index between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.
Change from Baseline of Lipid and Immune Profile measured in Blood | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of the lipid and immune profile of subjects treated with MERIVA® versus placebo. In particular, an omic-type approach will reveal alterations in lipid and energy metabolism, including lipoproteins, low molecular weight metabolites and individual lipid molecules, together with their degree of (poly) (non) saturation (blood panel including: leptin, adiponectin, Brain-derived Neurotrophic Factor, proinflammatory mediators such as Tumor Necrosis Factor alpha, interleukin-1 beta and interleukin-6, prostaglandins and reactive species of oxygen / nitrogen, inflammasome).
  The differences between genders are considered.
Change from Baseline of Brain-Derived Neurotrophic Factor (BDNF) and p66Shc Gene Expression measured in Blood | Change from Baseline (T0) to 6 months of treatment (T6).
  Evaluation in comparison to baseline of the lipid and immune profile of subjects treated with MERIVA® versus placebo. In particular, a sample of Peripheral Blood Mononuclear Cells (PBMC) will be separated for the measurement of the expression, by means of real-time Polymerase Chain Reaction (RT-PCR), of the neurotrophin Brain-Derived Neurotrophic Factor (BDNF) and of the p66Shc gene, which are involved in the response to lifestyle changes, including diets and exercise.
  The differences between genders are considered.
Rate and Characterization of Adverse Events occurred to Subjects | Pre-Screening (T-1) / Baseline (T0) / After 3 months of treatment (T3) / After 6 months of treatment (T6) / After 12 months of treatment (T12).
  Evaluation of the number, rate and characteristics of the adverse events occurring to subjects treated with MERIVA® versus placebo.
  The differences between genders are considered.

OTHER OUTCOMES:
Intestinal Microbiotic Profile Assessment in Stool Sample | Change from Baseline (T0) to 6 months of treatment (T6) and 12 months of treatment (T12).
  Evaluation in comparison to baseline of the intestinal microbiotic profile of subjects. Any differences between the groups treated with MERIVA® versus placebo will be recorded.
  The differences between genders are considered.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Giaccari, Prof., Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- S.C. di Endocrinologia e Diabetologia, Policlinico Universitario "Agostino Gemelli", Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen RC, Caracciolo B, Brayne C, Gauthier S, Jelic V, Fratiglioni L. Mild cognitive impairment: a concept in evolution. J Intern Med. 2014 Mar;275(3):214-28. doi: 10.1111/joim.12190. PMID 24605806
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Mrak RE, Griffin WS. Potential inflammatory biomarkers in Alzheimer's disease. J Alzheimers Dis. 2005 Mar;8(4):369-75. doi: 10.3233/jad-2005-8406. PMID 16556968
- [Background] Schrijvers EM, Witteman JC, Sijbrands EJ, Hofman A, Koudstaal PJ, Breteler MM. Insulin metabolism and the risk of Alzheimer disease: the Rotterdam Study. Neurology. 2010 Nov 30;75(22):1982-7. doi: 10.1212/WNL.0b013e3181ffe4f6. PMID 21115952
- [Background] Matsuzaki T, Sasaki K, Tanizaki Y, Hata J, Fujimi K, Matsui Y, Sekita A, Suzuki SO, Kanba S, Kiyohara Y, Iwaki T. Insulin resistance is associated with the pathology of Alzheimer disease: the Hisayama study. Neurology. 2010 Aug 31;75(9):764-70. doi: 10.1212/WNL.0b013e3181eee25f. Epub 2010 Aug 25. PMID 20739649
- [Background] Cicero AFG, Fogacci F, Morbini M, Colletti A, Bove M, Veronesi M, Giovannini M, Borghi C. Nutraceutical Effects on Glucose and Lipid Metabolism in Patients with Impaired Fasting Glucose: A Pilot, Double-Blind, Placebo-Controlled, Randomized Clinical Trial on a Combined Product. High Blood Press Cardiovasc Prev. 2017 Sep;24(3):283-288. doi: 10.1007/s40292-017-0206-3. Epub 2017 May 23. PMID 28537012
- [Background] Giugliano G, Salemme A, De Longis S, Perrotta M, D'Angelosante V, Landolfi A, Izzo R, Trimarco V. Effects of a new nutraceutical combination on cognitive function in hypertensive patients. Immun Ageing. 2018 Feb 7;15:7. doi: 10.1186/s12979-017-0113-4. eCollection 2018. PMID 29445414
- [Background] Cox KH, Pipingas A, Scholey AB. Investigation of the effects of solid lipid curcumin on cognition and mood in a healthy older population. J Psychopharmacol. 2015 May;29(5):642-51. doi: 10.1177/0269881114552744. Epub 2014 Oct 2. PMID 25277322
- [Background] Tabrizi R, Vakili S, Lankarani KB, Akbari M, Mirhosseini N, Ghayour-Mobarhan M, Ferns G, Karamali F, Karamali M, Taghizadeh M, Kouchaki E, Asemi Z. The Effects of Curcumin on Glycemic Control and Lipid Profiles Among Patients with Metabolic Syndrome and Related Disorders: A Systematic Review and Metaanalysis of Randomized Controlled Trials. Curr Pharm Des. 2018;24(27):3184-3199. doi: 10.2174/1381612824666180828162053. PMID 30156145
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Berry A, Cirulli F. The p66(Shc) gene paves the way for healthspan: evolutionary and mechanistic perspectives. Neurosci Biobehav Rev. 2013 Jun;37(5):790-802. doi: 10.1016/j.neubiorev.2013.03.005. Epub 2013 Mar 20. PMID 23524280
- [Background] Berry A, Bucci M, Raggi C, Eriksson JG, Guzzardi MA, Nuutila P, Huovinen V, Iozzo P, Cirulli F. Dynamic changes in p66Shc mRNA expression in peripheral blood mononuclear cells following resistance training intervention in old frail women born to obese mothers: a pilot study. Aging Clin Exp Res. 2018 Jul;30(7):871-876. doi: 10.1007/s40520-017-0834-4. Epub 2017 Sep 26. PMID 28952131
- See also: Sponsor company website — http://www.indena.com/